CLINICAL TRIAL: NCT06813196
Title: Forest Bathing Intervention for Persons Living with Dementia and Family Carers: a Feasibility Study
Brief Title: Forest Bathing Intervention for Persons Living with Dementia and Family Carers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Young Women's Christian Association (Other)
Responsible Party: Principal Investigator, Choy Chak Pui Jacky, Research Assistant Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EA240180
Record Dates: First submitted 2025-01-27; First posted 2025-02-06 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Dementia; Caregiver Mental Health
Keywords: Forest bathing
MeSH Terms: conditions — Dementia | interventions — Forest Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Forest bathing (Experimental): The modified forest bathing intervention was designed by a qualified forest therapist certified by the Association of Nature and Forest Therapy. The intervention protocol was developed based on existing forest bathing protocol and modified after field-testing with family caregivers. The intervention consisted of 3 sessions, delivered every two weeks, with approximately two hours per session. Each session took place at a suitable park in the participant's community. During the session, a group of 6 to 8 dyads of people living with dementia and their caregivers were guided by a trained forest therapy guide to engage in nature-based activities, such as walking in the woods, listening to the nature, and interacting with objects in the nature through different sensations. In between sessions, caregivers were encouraged to guide the PLwD and practice similar nature-based activities at times and locations at their convenience.
  Interventions: Behavioral: Forest Bathing
- Art activity (Active Comparator): The art activity intervention was modified from usual art activity session organised by the social service providers for family caregivers and PLwD. It consisted of 3 sessions, delivered every two weeks, with approximately two hours per session. Each session took place in an elderly community centre in the participant's neighbourhood. During the session, participants were guided to engage in individual or collaborative art activities of different forms, such as photo frame of dried flowers, plushball painting, and paper quilling. All the sessions were delivered by a social worker or program worker with experience in art-based activities.
  Interventions: Behavioral: Art activity

INTERVENTIONS:
Behavioral: Forest Bathing — Forest bathing intervention is a group structured psychosocial intervention. Its core therapeutic element is its nature-based activities that took place in an outdoor green space. During the session, participants would be guided by a trained forest therapy guide to engage in nature-based activities, such as walking in the woods, listening to the nature, and interacting with objects in the nature through different sensations.
  Arms: Forest bathing
Behavioral: Art activity — Art activity intervention is a group semi-structured psychosocial intervention. Its main therapeutic element is its engagement in art-based activites. During the session, participants would be guided in individual or collaborative art activities of different forms, such as painting, paper arts, and dried flower art, by an experienced interventionist in an activity room.
  Arms: Art activity

SUMMARY:
This study assessed the feasibility and acceptability of a forest bathing intervention for people living with dementia and their family carers, and examined its effectivness on care burden and quality of life by comparing to an art activty programme as control group.

ELIGIBILITY:
Inclusion Criteria:

* For family careivers:
* taking care of a family member living with dementia in the community,
* For people living with dementia:
* Clinical diagnosis of mild to moderate dementia

Exclusion Criteria:

* For both:
* Unable to communicate in Chinese or Cantonese
* Unable to participate meaningfully in group activities due to intellectual disability, visual impairment, hearing impairment, or other health conditions, were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2024-08-17 (Actual); Study Completion 2024-08-17 (Actual)

PRIMARY OUTCOMES:
Change in Caregiver's Care Burden measured by 12-item version of Zarit Burden Interview (ZBI-12) | Baseline and 6 weeks
  Possible range: 0-48, with higher scores indicate a worse outcome
Change in Caregiver's Depressive Symptoms measured by the Depression subscale of Hospital Anxiety and Depression Scale (HADS-D) | Baseline and 6 weeks
  Possible range: 0-21, with higher scores indicate a worse outcome
Change in Caregiver's Anxiety Symptoms measured by the Anxiety subscale of Hospital Anxiety and Depression Scale (HADS-A) | Baseline and 6 weeks
  Possible range: 0-21, with higher scores indicate a worse outcome

SECONDARY OUTCOMES:
Change in Caregiver's Positive Aspect of Caregiving measured by the Positive Aspect of Caregiving Scale (PACS) | Baseline and 6 weeks
  Possible range: 11-55, with higher scores indicate a better outcome
Change in Caregiver's Caregiving Self-Efficacy measured by the Revised Scale for Caregiving Self-Efficacy (CSE-R) | Baseline and 6 weeks
  Possible range: 0-100, with higher scores indicate a better outcome
Change in Caregiver's Health-related Quality of Life measured by the Visual Analogue Scale of EuroQol 5-dimension 5-level (EQ5D5L VAS) | Baseline and 6 weeks
  Possible range: 0-100, with higher scores indicate a better outcome
Change in Neuropsychiatric Symptoms of Person Living with Dementia measured by the Neuropsychiatric Inventory - Questionnaire (NPI-Q) | Baseline and 6 weeks
  Possible range: 0-12, with higher scores indicate a worse outcome
Change in Health-related Quality of Life of Person Living with Dementia measured by the Visual Analogue Scale of EuroQol 5-dimension 5-level (EQ5D5L VAS) | Baseline and 6 weeks
  Possible range: 0-100, with higher scores indicate a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Chak Pui Jacky Choy, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No